CLINICAL TRIAL: NCT03090230
Title: A Prospective, Multicenter, Non-Blinded, Non-Randomized Study of the RelayPro Thoracic Stent-Graft in Subjects With Traumatic Injury of the Descending Thoracic Aorta
Brief Title: Study of the Relay Pro® Thoracic Stent-Graft in Subjects With Traumatic Injury of the Descending Thoracic Aorta
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bolton Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IP-0018-16
Record Dates: First submitted 2017-03-07; First posted 2017-03-24 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-04

CONDITIONS: Other Specified Injury of Thoracic Aorta
Keywords: Descending Thoracic Aorta; DTA; Transection; Traumatic Injury of the Descending Thoracic Aorta

STUDY DESIGN:
Intervention Model Description: Subject must have a traumatic injury of the descending thoracic aorta that occurred no more than 30 days prior to the planned stent implant procedure. All subjects enrolled, will be included in the patient population for the primary analysis. All subjects implanted with the RelayPro Thoracic Stent-Graft will be included in the patient population for the secondary analyses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Relay Pro Thoracic Stent-Graft System (Experimental): The Relay Pro arm includes subjects who receive the device to treat traumatic injury of the descending thoracic aorta with the RelayPro Thoracic Stent-Graft System
  Interventions: Device: Relay Pro Thoracic Stent-Graft System

INTERVENTIONS:
Device: Relay Pro Thoracic Stent-Graft System — RelayPro Thoracic Stent-Grafts are designed for the management of patients with aneurysms and penetrating ulcers within the descending thoracic aorta (DTA). The device is designed specifically for use in the thoracic aorta.

SUMMARY:
The purpose of this study is to investigate the safety and effectiveness of the RelayPro Thoracic Stent-Grafts in subjects with traumatic injury of the descending thoracic aorta (DTA)

DETAILED DESCRIPTION:
This is a prospective, multicenter, non-blinded, non-randomized study of the RelayPro Thoracic Stent-Graft in subjects with traumatic injury of the DTA in subjects who are candidates for endovascular repair.The primary objective of the study is all-cause mortality at 30 days post procedure.

The secondary objectives of the trial will include descriptive analyses of procedural and post-procedural observations through 5 years of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Subject must have a traumatic injury of the descending thoracic aorta that occurred no more than 30 days prior to the planned stent implant procedure
* Proximal and distal landing zones with diameter between 19 mm and 42 mm.
* Subject must have a proximal attachment zone distal to the left common carotid and a distal attachment zone proximal to the origin of the celiac artery.
* The length of the attachment zones will depend on the intended stent graft diameter.

  1. The proximal attachment zone should be: i. 15 mm for 22 - 28 mm grafts with bare stent (20 mm for RelayPro grafts with non-bare stent). ii. 20 mm for 30 - 46 mm grafts with bare stent (25 mm for RelayPro grafts with non-bare stent).
  2. The distal attachment zone should be 20 mm for all Relay Pro grafts.
* Coverage of the left subclavian artery is permitted. Revascularization of the left subclavian artery may be considered in all cases by the treating physician and, especially, in anatomies where revascularization is determined to be clinically necessary
* Proximal and distal attachment zones containing a straight segment (non-tapered, non-reverse tapered, defined by <10% diameter change) with lengths equal to or greater than the required attachment length for the intended device.
* Adequate iliac or femoral artery access for introduction of the RelayPro delivery system. Alternative methods to gain proper access may be utilized (e.g., iliac conduit).
* Subject willing to comply with the follow-up evaluation schedule.
* Subject (or Legally Authorized Representative, LAR) agrees to sign an Informed Consent Form prior to treatment

Exclusion Criteria:

* Significant stenosis, calcification, thrombus, or tortuosity of intended fixation sites that would compromise fixation or seal of the device.
* Planned coverage of left carotid or celiac arteries; or anatomic variants that may compromise circulation to the carotid, vertebral, or innominate arteries after device placement, and are not amenable to subclavian revascularization
* Prior endovascular or surgical repair in the DTA. The device may not be placed within any prior endovascular or surgical graft.
* Concomitant aneurysm/disease of the ascending aorta, aortic arch, or abdominal, aorta requiring repair.
* Prior abdominal aortic aneurysm repair (endovascular or surgical) that was performed less than 6 months prior to the planned stent implant procedure.
* Untreatable allergy or sensitivity to contrast media or device components.
* Known or suspected connective tissue disorder.
* Blood coagulation disorder or bleeding diathesis for which the treatment cannot be suspended for one week pre- and/or post-repair.
* Coronary artery disease with unstable angina.
* Severe congestive heart failure (New York Heart Association functional class IV).
* Stroke and/or Myocardial Infarction within 3 months of the planned treatment date.
* Pulmonary disease requiring the routine (daily or nightly) need for oxygen therapy outside the hospital setting.
* Acute renal failure or chronic renal insufficiency, and not receiving dialysis.
* Hemodynamically unstable.
* Active systemic infection and/or mycotic aneurysms.
* Morbid obesity or other condition that may compromise or prevent the necessary imaging requirements.
* Injury Severity Score of 75.
* Less than two-year life expectancy.
* Current or planned participation in an investigational drug or device study that has not completed primary endpoint evaluation.
* Currently pregnant or planning to become pregnant during the course of the study.
* Medical, social, or psychological issues that Investigator believes may interfere with treatment or follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2025-11-22 (Estimated)

PRIMARY OUTCOMES:
Mortality post-procedure | 30 days
  All-cause mortality at 30 days post-procedure

SECONDARY OUTCOMES:
Successful device delivery and deployment | During Implantation
  Successful delivery and deployment of the device, including withdrawal of the delivery system, will be assessed with angiography during the index procedure at the Treatment Visit.
Loss of stent-graft patency | 1 month, 6 months, 12 months, and annually through 5 years
  Loss of stent-graft patency through 5 years
Aortic rupture | 1 month, 6 months, 12 months, and annually through 5 years
  Aortic rupture will be assessed at each follow-up visit with CT scans, or MRIs for subjects unable to tolerate contrast media
Stent fractures in the attachment zone | 1 month, 6 months, 12 months, and annually through 5 years
  Stent fractures in the attachment zone will be assessed at each follow-up visit with CT scans, or MRIs for subjects unable to tolerate contrast media
Endoleaks | 1 month, 6 months, 12 months, and annually through 5 years
  Persistence of blood flow outside the lumen of the stent-graft but within the native aorta or adjacent vascular segment being treated by the stent-graft
Compression of stent-graft | 1 month, 6 months, 12 months, and annually through 5 years
  Extra-luminal compression of the stent-graft will be assessed at each follow-up visit with xrays, CT scans, or MRIs for subjects unable to tolerate contrast media
Erosion and/or extrusion | 1 month, 6 months, 12 months, and annually through 5 years
  Erosion and extrusion will be assessed at each follow-up visit with CT scans, or MRIs for subjects unable to tolerate contrast media
Aortic expansion | 1 month, 6 months, 12 months, and annually through 5 years
  Aortic expansion (> 5mm) compared to the first post-procedural CT
Endograft infection | 1 month, 6 months, 12 months, and annually through 5 years
  Infection of stent-graft
Incidence of open or endovascular secondary interventions | 1 month, 6 months, 12 months, and annually through 5 years
  Incidence of open or endovascular secondary interventions to treat malperfusion, rupture, aneurysm formation, or aortic expansion
Migration | 1 month, 6 months, 12 months, and annually through 5 years
  Stent migration (> 10 mm) compared to the first post-procedural CT; formation, or aortic expansion
Major adverse events | 1 month, 6 months, 12 months, and annually through 5 years
  death, stroke, paralysis formation, or aortic expansion
Aortic-related death | 1 month, 6 months, 12 months, and annually through 5 years
  formation, or aortic expansion
Vascular access complications | During the initial implant attempt
  The Time Frame for reporting is during the Treatment Visit. Data should be captured upon conclusion of the Treatment Visit. Outcome measures include successful delivery and deployment of the device, as well as withdrawal of the delivery system
All-cause mortality | 1 month, 6 months, 12 months, and annually through 5 years
  All causes where subject death is the result of a serious and device- or procedure related adverse effect. Unrelated and accidental deaths, for example a subject death due to injuries sustained from a gunshot wound, would not be included in the evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Ben Starnes, MD, Principal Investigator — University of Washington; Ravi Rajani, MD, Principal Investigator — Emory University
Locations (16):
- United States (16):
  - University of California, Irvine, Irvine, California
  - Stanford Medicine, Stanford, California
  - Yale School of Medicine, New Haven, Connecticut
  - Grady Memorial Hospital, Atlanta, Georgia
  - Indiana University Health, Indianapolis, Indiana
  - University of Iowa Hospital and Clinic, Iowa City, Iowa
  - University of Maryland Medical Center, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center / Harvard Medical School, Boston, Massachusetts
  - St. Louis University, St Louis, Missouri
  - Atrium Health, Charlotte, North Carolina
  - University Hospitals, Cleveland, Ohio
  - University of Pennsylvania Medical Center / Penn Presbyterian, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Virginia, Charlottesville, Virginia
  - University of Washington, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No